CLINICAL TRIAL: NCT07227012
Title: AN INTERVENTIONAL OPEN-LABEL PHASE 1B/2 STUDY TO EVALUATE SAFETY, PHARMACOKINETICS, AND PRELIMINARY EFFICACY OF PF-08634404 AS MONOTHERAPY AND COMBINATION THERAPY IN ADULT PARTICIPANTS WITH UNRESECTABLE LOCALLY ADVANCED OR METASTATIC HEPATOCELLULAR CARCINOMA
Brief Title: A Study to Learn About Study Medicine Called PF-08634404 as a Single Treatment and Combination Treatment in Adult Participants With a Liver Cancer Called Hepatocellular Carcinoma, That is Too Advanced to be Removed by Surgery and May Have Spread to Other Parts of the Body.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C6461013; 2025-523525-17-00 (EU CTIS Number); Symbiotic-GI-13 (Other: Pfizer)
Record Dates: First submitted 2025-11-07; First posted 2025-11-12 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Carcinoma, Hepatocellular; Hepatocellular Cancer; Hepatocellular Carcinoma; Unresectable Hepatocellular Carcinoma; Liver Neoplasms; Advanced Hepatocellular Carcinoma; Metastatic Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Liver cancer; Liver Neoplasms
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Phase 1b (Experimental): Participants will be allocated to sequential dose levels of PF-08634404 and ipilimumab.
  Interventions: Biological: PF-08634404; Biological: Ipilimumab
- Phase 2 (Experimental): Participants will be randomized to receive either PF-08634404 monotherapy or PF-08634404 combined with ipilimumab.
  Interventions: Biological: PF-08634404; Biological: Ipilimumab

INTERVENTIONS:
Biological: PF-08634404 — Solution for infusion
Biological: Ipilimumab — Solution for infusion
  Other Names: YERVOY

SUMMARY:
The purpose of this study is to learn about the effects of study medicine (PF-08634404) when given alone or with another antibody (ipilimumab) for the treatment of a type of liver cancer called hepatocellular carcinoma (HCC) that is either locally advanced (spread to nearby tissues) or has spread to other parts of the body.

To join the study, participants must meet the following conditions:

* Be 18 years or older.
* Have locally advanced or metastatic HCC.
* Is not a candidate for complete surgical or loco-regional therapies.
* Have not received any whole-body treatment for HCC.

Participants will receive PF-08634404 either alone or in combination with ipilimumab. The medicine will be given through intravenous (IV) infusions, which means it will be administered directly into a vein. All treatments will take place at clinical trial sites, where trained medical staff will monitor participants during and after each visit.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at screening.
* Locally advanced or metastatic HCC with diagnosis confirmed by histology/cytology or clinically by AASLD criteria (for patients with cirrhosis). Participants without cirrhosis require histological confirmation of diagnosis.
* Disease that is not amenable to curative surgical and/or locoregional therapies, or progressive disease after surgical and/or locoregional therapies.
* At least 1 measurable (as defined by RECIST 1.1 per investigator) and untreated lesion.
* Adequate hepatic, liver, and renal function
* No prior systemic therapy for HCC.
* ECOG performance status 0 or 1
* Child-Pugh Class A

Key Exclusion Criteria:

* Moderate or severe ascites.
* History of hepatic encephalopathy.
* Participants with known active CNS lesions, including leptomeningeal metastasis, brainstem, meningeal, or spinal cord metastases or compression.
* Clinically significant risk of hemorrhage or fistula.
* Participants with any history of another malignancy within 3 years.
* History of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
* Participants with active autoimmune diseases requiring systemic treatment within the past 2 years.
* Clinically significant cardiovascular disease within 6 months prior to the first dose.
* Major surgery or severe trauma within 4 weeks prior to the first dose or planned major surgery during the study.
* History of severe bleeding tendency or coagulation dysfunction.
* History of severe ulcers, unhealed wounds, gastrointestinal perforation, abdominal fistula, gastrointestinal obstruction, intra-abdominal abscess, or acute gastrointestinal bleeding, including bleeding event due to esophageal and/or gastric varices, within 6 months prior to the first dose.
* Participants with acute, chronic or symptomatic infections.
* Participants with history of immunodeficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-10-18 (Estimated); Study Completion 2028-10-17 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events | Through end of study and up to approximately 24 months
  Adverse Events as characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), timing, seriousness, and relationship to study intervention.
Phase 1b: Number of participants with Dose limiting toxicities (DLT) | Through 90 days after the last dose of study intervention; Approximately 24 months
  DLTs are a predefined set of adverse events that are at least possibly related to any or all of the study interventions. The number of participants who experienced DLTs during the DLT observation period.
Phase 2: Confirmed Overall Response Rate (ORR) using RECIST 1.1 as assessed by investigator | Approximately 24 months
  ORR is the proportion of participants with a best overall response (BOR) of confirmed CR or confirmed PR per RECIST 1.1 by investigator.
Phase 2: Recommended dose of PF-08634404 in combination with ipilimumab | Approximately 24 months
  The doses of PF-08634404 and ipilimumab selected to be used in combination based on safety, tolerability, pharmacokinetics, and initial anti-tumor efficacy from Phase 2.

SECONDARY OUTCOMES:
Phase 1b: Confirmed Objective Response Rate (ORR) using RECIST 1.1 as assessed by investigator | Approximately 24 months
  ORR is the proportion of participants with a best overall response of confirmed Complete Response (CR) or confirmed Partial Response (PR) per RECIST 1.1 by investigator.
Duration of Response (DOR) per RECIST 1.1 by investigator | Approximately 24 months
  DOR is the time from the first documentation of objective response (CR or PR that is subsequently confirmed) to the date of first documented disease progression per RECIST 1.1 as assessed by investigator, or death due to any cause, whichever occurs first.
Progression Free Survival (PFS) per RECIST 1.1 by investigator | Approximately 24 months
  PFS is defined as the time from the date of first dose to the date of first documented disease progression per RECIST 1.1 as assessed by investigator, or death due to any cause, whichever occurs first.
Overall Survival (OS) | Approximately 24 months
  OS is defined as the time from the date of first dose to the date of death due to any cause.
Number of Participants With Clinical Laboratory Abnormalities | Time from the date of first dose of study intervention through 30-37 days after last dose of study intervention (assessed up to approximately 24 months)
  Laboratory abnormalities as characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), and timing
Pharmacokinetics (PK): Serum concentrations of PF-08634404 | Up to 24 months
  Predose and/or postdose concentrations of PF-08634404 in combination with ipilimumab.
Incidence of antidrug antibody against PF-08634404 | Up to 24 months
  To evaluate immunogenicity of PF-08634404 in combination with ipilimumab.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pan American Center for Oncology Trials, LLC, San Juan, Other, Puerto Rico

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C6461013